CLINICAL TRIAL: NCT01409200
Title: Pre-Surgical Androgen Deprivation Therapy With or Without Axitinib in Previously Untreated Prostate Cancer Patients With Known or Suspected Lymph Node Metastasis
Brief Title: Antiandrogen Therapy With or Without Axitinib Before Surgery in Treating Patients With Previously Untreated Prostate Cancer With Known or Suspected Lymph Node Metastasis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0231; NCI-2015-01711 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2011-02749; 2011-0231 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Malignant Neoplasm in Lymph Node; Prostate Ductal Adenocarcinoma; Stage III Prostate Adenocarcinoma AJCC v7; Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: conditions — Lymphatic Metastasis | interventions — Androgen Antagonists; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (antiandrogen therapy, axitinib, surgery) (Experimental): Patients receive antiandrogen therapy per standard care and axitinib PO BID for 4 months. Patients then undergo radical prostatectomy and pelvic lymph node dissection.
  Interventions: Drug: Antiandrogen Therapy; Drug: Axitinib; Procedure: Radical Prostatectomy; Procedure: Regional Lymph Node Dissection
- Arm II (antiandrogen therapy, surgery) (Active Comparator): Patients receive antiandrogen therapy per standard care for 4 months and then undergo radical prostatectomy and pelvic lymph node dissection.
  Interventions: Drug: Antiandrogen Therapy; Procedure: Radical Prostatectomy; Procedure: Regional Lymph Node Dissection

INTERVENTIONS:
Drug: Antiandrogen Therapy — Given per standard of care
  Other Names: ADT; Androgen Deprivation Therapy; Anti-androgen Therapy; Anti-androgen Treatment; Antiandrogen Treatment; Hormone Deprivation Therapy; Hormone-Deprivation Therapy
Drug: Axitinib — Given PO
  Other Names: AG-013736; AG013736; Inlyta
  Arms: Arm I (antiandrogen therapy, axitinib, surgery)
Procedure: Radical Prostatectomy — Undergo radical prostatectomy
  Other Names: Prostatovesiculectomy
Procedure: Regional Lymph Node Dissection — Undergo pelvic lymph node dissection

SUMMARY:
This randomized phase IIA trial studies how well antiandrogen therapy works with or without axitinib before surgery in treating patients with previously untreated prostate cancer that is known or suspected to have spread to lymph nodes. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as antiandrogen therapy may lessen the amount of androgen made by the body. Axitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known if antiandrogen therapy is more effective with or without axitinib before surgery in treating patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the proportion of patients progression-free one year after treatment with axitinib plus androgen deprivation versus (vs.) androgen deprivation therapy alone and surgery in newly diagnosed prostate cancer patients with lymph node metastases (TxN1M0 or TxNxM1a) or clinical suspicion of lymph node metastases.

SECONDARY OBJECTIVES:

I. To compare the rate of pathologic complete response (pCR) in the primary tumor.

II. To evaluate time to progression. III. Describe the perioperative and postoperative morbidity of pre-surgical treatment.

IV. Evaluate the effects of a 6-month time course of androgen deprivation with or without axitinib in prostate cancer tissue and blood.

V. Develop a prospective tissue archive of prostate tumors that have metastasized to lymph nodes.

OUTLINE:

Patients receive antiandrogen therapy per standard care for 8 weeks.

Patients are then randomized to 1 of 2 treatment arms.

ARM I: Patients receive antiandrogen therapy per standard care and axitinib orally (PO) twice daily (BID) for 4 months. Patients then undergo radical prostatectomy and pelvic lymph node dissection.

ARM II: Patients receive antiandrogen therapy per standard care for 4 months and then undergo radical prostatectomy and pelvic lymph node dissection.

After completion of study treatment, patients are followed up at 1 and 3 months, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adenocarcinoma of the prostate that in the opinion of the urologist could be resected after response to systemic therapy; ductal adenocarcinoma is permitted
* Patients must be regarded as acceptable surgical risk for radical prostatectomy and confirm their intention to undergo radical prostatectomy at the end of the pre-surgical therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 2 or better
* All patients must have thorough tumor staging and meet at least one of the following criteria:

  * Either lymph node biopsy or lymph node dissection demonstrating lymph node metastasis by prostate cancer
  * Non-bulky (< 5 cm) regional pelvic or distant lymphadenopathy visualized on computed tomography (CT)/magnetic resonance imaging (MRI) scan; lymph node biopsy is required if < 2.0 cm or in atypical distribution
  * Primary tumor Gleason score >= 8 and serum prostate-specific antigen (PSA) concentration >= 25 ng/mL, indicating high risk of occult lymph node metastases
  * Primary clinical tumor stage of T3 and Gleason score >= 7, indicating high risk of occult lymph node metastases
  * Primary tumor stage T4, indicating high risk of occult lymph node metastases; patients in any of these groups and less than 3 sites of non-predominantly lytic bone metastasis will be still considered eligible for the trial; the 2010 American Joint Committee on Cancer (AJCC) staging system will be followed
* Prior hormonal therapy (luteinizing hormone-releasing hormone [LHRH] agonist/antagonist with or without antiandrogen) up to 8 weeks is permitted
* Absolute peripheral neutrophil count (ANC) of >= 1,500/mm^3
* Platelet count of >= 100,000/mm^3
* Total bilirubin of =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN
* Serum creatinine =< 1.5 x ULN or clearance >= 60 mL/min (measured or calculated)
* Urinary protein < 2+ by urine dipstick (if >= 2+, a 24-hour urine protein must show protein < 2 g per 24 hours)
* Patients or their partners must be surgically sterile or must agree to use effective contraception while receiving study treatment and for at least 3 months thereafter; the definition of effective contraception should be in agreement with local regulation and based on the judgment of the principal investigator or a designated associate
* Patients must sign the current institutional review board (IRB) approved informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of the institution, and willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* All patients must have a surgical and medical oncology consult prior to signing informed consent

Exclusion Criteria:

* Patients with biopsy-proven small cell or sarcomatoid histology
* Patients with clinical or radiological evidence of bone (>= 3 sites, or predominantly lytic if < 3) or other extranodal metastasis
* Patients who have had prior chemotherapy, experimental agents for prostate cancer, or patients receiving more than 8 weeks of prior hormone therapy will be excluded
* Gastrointestinal abnormalities such as inability to take oral medication; requirement for intravenous alimentation; prior surgical procedures affecting absorption including total gastric resection; treatment for active peptic ulcer disease in the past 6 months; active gastrointestinal bleeding as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy; malabsorption syndromes
* Anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors (i.e., verapamil, ketoconazole, miconazole, itraconazole, erythromycin, telithromycin, clarithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir and delavirdine); grapefruit juice is also a CYP3A4 inhibitor
* Anticipated need for treatment with drugs that are known CYP3A4 or CYP1A2 inducers (i.e. carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort)
* Patients with any infectious process that, in the opinion of the investigator, could worsen or its outcome be affected as a result of the investigational therapy
* Patients with symptomatic congestive heart failure, unstable angina or myocardial infarction, coronary/peripheral artery bypass graft or repair, cerebrovascular accident or transient ischemic attack in the 12 months prior to randomization; or deep vein thrombosis or pulmonary embolism in the 6 months prior to randomization
* Persistently uncontrolled diabetes mellitus, oxygen-dependent lung disease, chronic liver disease, or human immunodeficiency virus (HIV) infection
* Inadequately controlled hypertension (defined as systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg) despite antihypertensive medication, or prior history of hypertensive crisis or hypertensive encephalopathy
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Anticipation of need for major surgical procedure during the course of the study other than as outlined by the protocol
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to randomization
* Serious, non-healing wound, active ulcer, or untreated bone fracture; any bone fractures must be healed
* Known hypersensitivity to any component of axitinib or prior use of axitinib
* Second malignancies (excluding non-melanoma skin cancer) unless treated with curative intent and disease-free for 3 years
* Overt psychosis, mental disability, otherwise incompetent to give informed consent, or history of non-compliance
* Planned participation in any other experimental drug study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-03-26 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Participants Progression-free 12 months after surgery | 12 months after surgery
  Time to Prostate-specific antigen (PSA)-progression measured from the date of radical prostatectomy to the occurrence of a serum PSA >1.0 ng/mL (confirmed by a second measurement at least 2 weeks apart). PSA-monitoring every 3 months after surgery for the first 12 months, every 4 months in the second year, every 6 months in the third to fifth year, and yearly thereafter until PSA or radiologic progression.

CONTACTS AND LOCATIONS:
Overall Officials: Amado J Zurita Saavedra, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org